CLINICAL TRIAL: NCT07175441
Title: A Phase 2a, Multicenter, Randomized, Open-Label Study to Assess the Efficacy, Safety, and Tolerability of RBS2418 in Combination With Tremelimumab Plus Durvalumab for Participants With Advanced Unresectable Hepatocellular Carcinoma
Brief Title: Evaluation of RBS2418 in Combination With Tremelimumab Plus Durvalumab in Participants With Advanced Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Riboscience, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBS2418-2002
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Unresectable Hepatocellular Carcinoma
Keywords: Advanced Unresectable Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: RBS2418, 200mg BID, plus STRIDE (Active Comparator): RBS2418 200 mg PO, BID in combination with STRIDE regimen
  Interventions: Drug: RBS2418; Drug: STRIDE (durvalumab + tremelimumab)
- Arm B: RBS2418, 800mg BID, plus STRIDE (Active Comparator): RBS2418 800 mg PO, BID in combination with STRIDE regimen
  Interventions: Drug: RBS2418; Drug: STRIDE (durvalumab + tremelimumab)
- Arm C: STRIDE alone (control) (Active Comparator): STRIDE regimen
  Interventions: Drug: STRIDE (durvalumab + tremelimumab)

INTERVENTIONS:
Drug: RBS2418 — RBS2418 is a specific immune modulator that works through the inhibition of ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1) and is designed to lead to anti-tumor immunity by protecting endogenous 2'-3'-cyclic guanosine monophosphate-adenosine monophosphate (cGAMP) from hydrolysis and leading to the activation of antigen-presenting cells followed by T cell activation.
  Arms: Arm A: RBS2418, 200mg BID, plus STRIDE; Arm B: RBS2418, 800mg BID, plus STRIDE
Drug: STRIDE (durvalumab + tremelimumab) — STRIDE: Tremelimumab 300 mg IV (Cycle 1 Day 1 only) Plus Durvalumab 1500 mg IV every 4 weeks

SUMMARY:
RBS2418 is a targeted immune modulator that inhibits ectonucleotide pyrophosphatase/phosphodiesterase 1 (ENPP1). It is designed to promote anti-tumor immunity by preserving endogenous 2'-3' cyclic guanosine monophosphate-adenosine monophosphate (cGAMP) from hydrolysis, thereby activating antigen-presenting cells and promoting robust T cell activation. Ideally, RBS2418 acts synergistically with CTLA-4 inhibitors, such as those in the STRIDE regimen (Tremelimumab plus Durvalumab). The hypothesis is that RBS2418 combined with STRIDE will be safe, well-tolerated, highly immunogenic, and enhance anti-tumor responses in adult participants with advanced, unresectable hepatocellular carcinoma (HCC) compared to STRIDE alone.

DETAILED DESCRIPTION:
In this Phase 2a study, participants must have advanced, unresectable HCC confirmed by radiology, histology or cytology. Participants must be eligible to receive the STRIDE regimen as first line therapy. Participants must have measurable disease per RECIST 1.1, an Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1 or 2, and predicted life expectancy of at least 12 weeks.

Up to approximately 220 participants will be enrolled and will receive therapy as part of their respective treatment group. Participants will receive study treatment of RBS2418 at two different dose levels (200mg and 800mg) twice daily in combination with STRIDE or STRIDE alone with a treatment period consisting of 28-day cycles up to two years or until there is progressive disease, death, withdrawal, or study completion, whichever comes first.

Adverse Events (AEs) will be monitored throughout the study and graded in severity according to the guidelines outlined in the NCI CTCAE v5.0. AEs will be collected until up to 30 days after the last dose of RBS2418 or until resolution, whichever comes first. SAEs will be collected for 90 days after the last dose of RBS2418, or if the participant initiates new anti-cancer therapy, then 30 days after the RBS2418 last dose, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of signing informed consent.
2. Male and female participants with advanced, unresectable HCC who are eligible to receive STRIDE regimen as first line therapy.
3. Willing to submit a pre-treatment tissue sample (archival or fresh tissue if archival is not available).

Exclusion Criteria:

1. BCLC stage D disease at the time of screening or prior to first dose of RBS2418.
2. Child-Pugh class equal or higher than B8 at the time of screening or within 7 days prior to the first dose of study treatment.
3. Eligible for curative treatments (e.g., surgical resection, liver transplantation, or local ablation).
4. Evidence of rapid progression on prior therapy resulting in rapid clinical deterioration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From randomization until the first radiographic documentation of objective progression or death from any cause, assessed up to 2 years.
  Time in months from randomization until the first radiographic documentation of objective progression, as assessed using RECIST 1.1, or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death from any cause, assessed up to 2 years.
  Time in months from the date of randomization to the date of death from any cause.
Overall Response Rate (ORR) by RECIST 1.1 | From randomization to initial response, assessed up to 2 years
  ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) during the study using RECIST 1.1, among those with measurable disease.
Duration of Response (DOR) by RECIST 1.1 | From initial response to disease progression or death, assessed up to 2 years
  DOR is defined as time from initial response to disease progression or death.
Disease Control Rate (DCR) | From randomization to end of treatment or disease progression, assessed up to 2 years.
  DCR is defined as the percentage of participants who achieve a complete response (CR), partial response (PR) or stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - START Dallas Fort Worth, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No